CLINICAL TRIAL: NCT02467218
Title: Hyperbaric Oxygen Therapy in Fibromyalgia : Effect on Global Function
Brief Title: HBOT in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-7888-A
Record Dates: First submitted 2015-04-20; First posted 2015-06-09 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Hyperbaric Oxygen Treatment; Fibromyalgia; Global Function; Sleep; Chronic Pain; Depression; Anxiety
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Hyperbaric Oxygen Treatment (Experimental): If a participant is randomized to the group receiving the intervention, the participant will be receiving a baseline assessment functional magnetic resonance imaging (fMRI) and subsequently receiving hyperbaric oxygen treatment for 90 minutes, once daily, five times a week for 8 consecutive weeks (40 treatments with 100% oxygen at 2.0 ATA). A follow-up fMRI will be performed after the last day of treatment.
  Interventions: Other: Hyperbaric Oxygen Treatment
- Delayed Hyperbaric Oxygen Treatment (Experimental): If the participant is assigned to the cross group, the participant will also receive a baseline assessment functional magnetic resonance imaging (fMRI). However, it will be followed-up in a controlled manner for 3 months. After 3 months, the participant will be receiving hyperbaric oxygen treatment identical to Group A and a follow-up fMRI will be performed after the last treatment.
  Interventions: Other: Hyperbaric Oxygen Treatment

INTERVENTIONS:
Other: Hyperbaric Oxygen Treatment — Baseline and follow up fMRI and Oxygen treatment, 90 minutes, once daily, five times a week for 8 consecutive weeks in the hyperbaric chamber (40 treatments with 100% oxygen at 2.0 ATA)

SUMMARY:
Fibromyalgia (FM) is a chronic pain condition affecting several millions of Canadians. Although the etiology and pathophysiology are poorly understood, there is a well-recognized association between muscular pain in fibromyalgia and muscular hypoperfusion, hypoxia, abnormal muscle metabolism and oxidative stress. Currently there is no cure for FM. Pharmacological and non-pharmacological strategies are directed to control symptoms such as pain, fatigue, non-restorative sleep and depression.

Hyperbaric oxygen therapy (HBOT) is an intermittent inhalation of 100% oxygen in a hyperbaric chamber at a pressure higher than 1 absolute atmosphere. Physiological effect of HBOT is based on a dramatic increase in the amount of dissolved oxygen carried by the blood which enables oxygenation of ischemic areas with compromised circulation. It also activates oxidant-antioxidant system, stimulates angio- and neurogenesis, modulates inflammatory response, induces brain neuroplasticity and possesses analgesic effect.

While some interventions offer benefit for some patients, additional treatment alternatives are needed for patients with FM in whom currently available options are either ineffective or poorly tolerated. Given its physiological effect, HBOT could be considered as a potential therapy for treatment of underlying muscular hypoxia, optimizing oxidant- antioxidant system and controlling FM symptoms. The results from this study could therefore provide new information supporting the basic science underling the pathophysiology of this disease and stimulate novel therapies for patients suffering with FM.

ELIGIBILITY:
Inclusion Criteria:

* Function Improvement Questionnaire (Revised) score ≥ 60 during the baseline assessment.

Exclusion Criteria:

* Women with positive pregnancy test or plans to become pregnant during the study period
* Claustrophobia
* Seizure disorder
* Active asthma
* Severe chronic obstructive pulmonary disease
* Previous thoracic surgery
* History of pneumothorax
* History of severe congestive heart failure with left ventricular ejection fraction < 30%
* Unstable angina
* Chronic sinusitis
* Chronic or acute otitis media or major ear drum trauma
* Current treatment with bleomycin, cisplatin, doxorubicin and disulfiram
* Participation in another investigative drug or device trial currently or within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants finishing the study protocol | 3 months post treatment
  Feasibility as a number of participants finishing the study protocol
Number of participants experiencing intervention related adverse events | Start of Treatment to post 3 months
  Safety as a proportion of patients experiencing intervention-related adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Curtis K, Katz J, Djaiani C, O'Leary G, Uehling J, Carroll J, Santa Mina D, Clarke H, Gofeld M, Katznelson R. Evaluation of a Hyperbaric Oxygen Therapy Intervention in Individuals with Fibromyalgia. Pain Med. 2021 Jun 4;22(6):1324-1332. doi: 10.1093/pm/pnaa416. PMID 33594439